CLINICAL TRIAL: NCT01119950
Title: A Randomized, Double-blind, Placebo-controlled, 2-period, Cross-over Study to Assess the Efficacy and Safety of Differing Doses of NVA237 Administered Either Once Daily or Twice Daily, in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of NVA237 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2208; 2009-014038-11 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- NVA237 12.5 µg q.d. (Experimental): NVA237 12.5 µg once daily
  Interventions: Drug: NVA237 12.5 µg once daily
- NVA237 25.0 µg q.d. (Experimental): NVA237 25.0 µg once daily
  Interventions: Drug: NVA237 25.0 µg once daily
- NVA237 12.5 µg b.i.d. (Experimental): NVA237 12.5 µg twice daily
  Interventions: Drug: NVA237 12.5 µg twice daily
- NVA237 50.0 µg q.d. (Experimental): NVA237 50.0 µg once daily
  Interventions: Drug: NVA237 50.0 µg once daily
- NVA237 25.0 µg b.i.d. (Experimental): NVA237 25.0 µg twice daily
  Interventions: Drug: NVA237 25.0 µg twice daily
- NVA237 100.0 µg q.d. (Experimental): NVA237 100.0 µg once daily
  Interventions: Drug: NVA237 100.0 µg once daily
- NVA237 50.0 µg b.i.d. (Experimental): NVA237 50.0 µg twice daily
  Interventions: Drug: NVA237 50.0 µg twice daily
- Placebo (Placebo Comparator): Placebo to NVA237 once daily
  Interventions: Drug: Placebo to NVA237 once daily

INTERVENTIONS:
Drug: NVA237 12.5 µg once daily — NVA237 12.5 µg via dry powder inhaler once daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 12.5 µg q.d.
Drug: NVA237 25.0 µg once daily — NVA237 25.0 µg via dry powder inhaler once daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 25.0 µg q.d.
Drug: NVA237 12.5 µg twice daily — NVA237 12.5 µg via dry powder inhaler twice daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 12.5 µg b.i.d.
Drug: NVA237 50.0 µg once daily — NVA237 50.0 µg via dry powder inhaler once daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 50.0 µg q.d.
Drug: NVA237 25.0 µg twice daily — NVA237 25.0 µg via dry powder inhaler twice daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 25.0 µg b.i.d.
Drug: NVA237 100.0 µg once daily — NVA237 100.0 µg via dry powder inhaler once daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 100.0 µg q.d.
Drug: NVA237 50.0 µg twice daily — NVA237 50.0 µg via dry powder inhaler twice daily for 28 days during either period 1 or during period 2.
  Arms: NVA237 50.0 µg b.i.d.
Drug: Placebo to NVA237 once daily — Placebo to NVA237 via dry powder inhaler once daily for 28 days during either period 1 or during period 2.
  Arms: Placebo

SUMMARY:
This study was designed to investigate the efficacy and safety of NVA237, a long-acting muscarinic antagonist, in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 40 years or more
* Diagnosis of Chronic Obstructive Lung Disease (COPD) (moderate to severe as classified by the Global Initiative for COPD (GOLD) Guidelines, 2008
* Smoking history of at least 10 pack-years
* Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) <80% and ≥30% of the predicted normal value
* Post-bronchodilator FEV1/Forced Vital Capacity (FVC) <0.7
* Symptomatic patients, according to daily electronic diary data between visit 2 (Day -8) and Visit 3 (Day 1), with a total score of 1 or more on at least 4 of the last 7 days prior to visit 3

Exclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization in the 6 weeks prior to the first visit
* Patients who have had a respiratory tract infection within 4 weeks prior to the first visit
* Patients with concomitant pulmonary disease
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions
* Patients with a history of asthma or a blood eosinophil count >600/mm3 or onset of symptoms prior to 40 years
* Patients with eczema, known high IgE levels or a known positive skin prick test
* Patients participating in the active phase of a pulmonary rehabilitation programme
* Patients contraindicated for the treatment with anticholinergics, long and short-acting beta-2 agonists or sympathomimetic amines
* Patients with a history of alpha-1 anti-trypsin deficiency
* Patients on long term oxygen therapy (>15hr per day)
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (6):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Belgium (3):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Genk
  - Novartis Investigative site, Jambes
- Novartis Investigative Site, München, Germany
- Hungary (6):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Törökbálint
- Netherlands (7):
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Helmond
  - Novartis Investigative Site, Veldhoven
  - Novartis Investigative Site, Zutphen
- Poland (3):
  - Novartis Investigative Site, Izabelin
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
- Spain (3):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Ponferrada

REFERENCES:
- [Derived] Arievich H, Overend T, Renard D, Gibbs M, Alagappan V, Looby M, Banerji D. A novel model-based approach for dose determination of glycopyrronium bromide in COPD. BMC Pulm Med. 2012 Dec 8;12:74. doi: 10.1186/1471-2466-12-74. PMID 23217058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to 1 of 8 treatment groups during period 1; participants were then switched to a different treatment group during period 2 after a 7 days wash out. Each period lasted up to 29 days.
Pre-assignment Details: For this crossover study, a participant is counted in 2 treatment groups
Groups:
- Overall Study: For the overall study, 388 participants were randomized and 1 non-randomized participant received drug in error and was discontinued. This participant was excluded from randomized number of patients but included in number of treated participants and in the safety set.
  Out of the 388 participants randomized, 341 completed study treatment and 47 discontinued, including 3 misrandomized participants who did not receive any study medication.
Period: Overall Study
Arm/Group | Overall Study
Started | 388 (These participants were randomized to 2 different treatment sequences during period 1 and 2.)
NVA237 12.5 ug q.d. | 96 (5 randomized and 2 misrandomized patients did not receive study drug, 80 completed, 9 discontinued.)
NVA237 25 ug q.d. | 99 (3 randomized participants did not receive study drug, 91 completed treatment, 5 discontinued.)
NVA237 12.5 ug b.i.d. | 99 (4 randomized participants did not receive study drug, 93 completed treatment, 2 discontinued.)
NVA237 50 ug q.d. | 96 (4 randomized participants did not receive study drug, 89 completed treatment, 3 discontinued.)
NVA237 25 ug b.i.d. | 100 (4 randomized participants did not receive study drug, 89 completed treatment, 7 discontinued.)
NVA237 100 ug q.d. | 98 (2 randomized participants did not receive study drug, 92 completed treatment, 4 discontinued.)
NVA237 50 ug b.i.d. | 94 (6 randomized and 1 misrandomized patients did not receive study drug, 82 completed, 5 discontinued.)
Placebo | 94 (3 randomized participants did not receive study drug, 82 completed treatment, 5 discontinued.)
Completed | 341 (These participants completed both periods 1 and 2)
Not Completed | 47
Not completed — Adverse Event | 25
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 4
Not completed — Administrative | 2
Not completed — Abnormal lab value | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Baseline/demographic measures are based on safety set
Groups:
- All Participants: All participants in the safety set
Arm/Group | All Participants
Number analyzed (Participants) | 386
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251
  Male | 135

OUTCOME MEASURES:

1. Secondary Outcome: Trough Forced Expiratory Volume in One Second for Once and Twice Daily Regimens of NVA237 for the Same Total Daily Dose of NVA237
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  FEV1 was measured between dosing regimens (over the range 20 micrograms to 55 micrograms total daily dose) after 28 days of treatment.
  Mean trough FEV1 was measured in response to all doses administered (12.5 µg q.d., 25.0 µg q.d., 12.5 µg b.i.d., 50 µg q.d., 25 µg b.i.d., 100 µg q.d., 50.0 µg b.i.d., and Placebo; see Outcome Measure # 19), and was used to compute modeled dose-response curves for once-daily and twice-daily regimens separately. The difference between those curves was computed at pre-specified theoretical doses (20 µg, 25 µg, 30 µg, 35 µg, 40 µg, 45 µg, 50 µg, and 55 µg) chosen at points likely to show the largest differences between the once-daily and twice-daily regimens. The theoretical responses to each dosing schedule separately and the difference between the once-daily and twice-daily regimens are represented below.
Time Frame: day 28
Population: Full analysis set includes all randomized patients who received at least one dose of study drug and data available for analysis. Only patients with non-missing values were included.
Measure: Mean (90% Confidence Interval); unit: Liters
Groups:
- Overall Study: A statistical modeling process was used to achieve the key objective. A set of 4 candidate models based on the Emax dose-response shape was derived plus their sigmoidal Emax counterparts (a total of 8 models) that describe the evolution of dose response over time. A model-averaging process was then employed to obtain response predictions as the weighted average of individual model predictions and confidence limits derived using a simulation-based procedure.
Arm/Group | Overall Study
Number analyzed (Participants) | 385
Liters
  Total daily dose 20 ug | 0.037 [0.013 to 0.053]
  Total daily dose 25 ug | 0.037 [0.013 to 0.052]
  Total daily dose 30 ug | 0.036 [0.013 to 0.051]
  Total daily dose 35 ug | 0.035 [0.013 to 0.050]
  Total daily dose 40 ug | 0.034 [0.013 to 0.049]
  Total daily dose 45 ug | 0.033 [0.013 to 0.047]
  Total daily dose 50 ug | 0.032 [0.012 to 0.046]
  Total daily dose 55 ug | 0.031 [0.012 to 0.045]

2. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second Area Under the Curve 0-24 Hours at Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-24 hours at day 28 of treatment was calculated from measurements taken at 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28.
  AUC FEV1 was measured in response to all doses administered (see Outcome Measure #20). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response * hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 82 | 90 | 91 | 90 | 92 | 91 | 82
Percentage of maximal response * hours | 28.9 [18.7 to 41.6] | 44.8 [31.6 to 58.8] | 49.0 [34.1 to 64.1] | 61.9 [48.0 to 74.0] | 65.7 [50.9 to 78.1] | 76.4 [64.8 to 85.1] | 79.3 [67.5 to 87.7]

3. Secondary Outcome: Forced Expiratory Volume in One Second AUC 0-24 Hours for Once and Twice Daily Regimens of NVA237 for the Same Total Daily Dose of NVA237, After 28 Days of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  The Area Under the Curve (AUC) 0-24 hours FEV1 between dosing regimens over the range 20 micrograms to 55 micrograms total daily dose at -25 min,-15 min (predose); 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28.
  AUC 0-24 hours FEV1 was measured in response to all doses administered (12.5 µg q.d., 25.0 µg q.d., 12.5 µg b.i.d., 50 µg q.d., 25 µg b.i.d., 100 µg q.d., 50.0 µg b.i.d., and Placebo; see Outcome Measure # 20), and was used to compute modeled dose-response curves for once-daily and twice-daily regimens separately. The difference between those curves was computed at pre-specified theoretical doses (20 µg, 25 µg, 30 µg, 35 µg, 40 µg, 45 µg, 50 µg, and 55 µg) chosen at points likely to show the largest differences between the once-daily and twice-daily regimens.
Time Frame: -25 min,-15 min (predose); 5 min,15 min, 1,2,3,4,6,8,10 hours, 11 hours 55min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Overall Study
Number analyzed (Participants) | 385
Liters
  Total daily dose 20 ug | 0.008 [-0.008 to 0.023]
  Total daily dose 25 ug | 0.008 [-0.008 to 0.024]
  Total daily dose 30 ug | 0.008 [-0.008 to 0.024]
  Total daily dose 35 ug | 0.008 [-0.008 to 0.023]
  Total daily dose 40 ug | 0.008 [-0.008 to 0.023]
  Total daily dose 45 ug | 0.008 [-0.008 to 0.022]
  Total daily dose 50 ug | 0.008 [-0.008 to 0.022]
  Total daily dose 55 ug | 0.007 [-0.007 to 0.021]

4. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second Area Under the Curve at Different Time Points (0-4 Hours, 0-8 Hours, 0-12 Hours, 12-24 Hours) on Day 28
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-4 Hours, 0-8 Hours, 0-12 Hours, 12-24 Hours were calculated from measurements taken at: 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28.
  AUC FEV1 was measured in response to all doses administered (see Outcome Measure #21). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 5 min,15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 82 | 90 | 91 | 90 | 92 | 91 | 82
Percentage of maximal response* hours
  AUC 0-4h (n=82,90,91,89,92,91,82) | 50.8 [38.7 to 63.6] | 66.9 [53.7 to 77.7] | 58.9 [45.9 to 71.5] | 79.7 [67.4 to 87.4] | 73.7 [60.6 to 83.4] | 88.3 [77.8 to 93.3] | 84.4 [73.0 to 91.0]
  AUC 0-8h (n=82,90,91,90,92,91,82) | 45.8 [33.2 to 58.8] | 62.8 [49.9 to 74.1] | 55.5 [42.0 to 68.4] | 77.1 [66.6 to 85.1] | 71.4 [59.1 to 81.2] | 87.1 [79.9 to 91.9] | 83.3 [74.3 to 89.7]
  AUC 0-12h (n=82,90,91,90,92,91,82) | 41.1 [28.8 to 54.5] | 58.3 [44.7 to 70.6] | 50.5 [37.0 to 64.1] | 73.6 [61.8 to 82.8] | 67.1 [54.0 to 78.1] | 84.8 [76.4 to 90.6] | 80.3 [70.1 to 87.7]
  AUC 12-24h (n=82,90,91,89,92,91,81) | 25.6 [15.5 to 42.5] | 40.1 [24.2 to 59.6] | 56.6 [31.4 to 78.2] | 56.4 [33.0 to 74.7] | 71.4 [41.5 to 87.8] | 71.2 [42.6 to 85.5] | 82.4 [51.2 to 93.5]

5. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second at 12 Hours at Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response within different doses/regimens of NVA237 was measured using FEV1 at 12 hours on day 28 of treatment.
  FEV1 was measured in response to all doses administered (see Outcome Measure #22). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 12 hours on day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 79 | 88 | 91 | 85 | 87 | 88 | 78
Percentage of maximal response | 27.1 [14.7 to 44.6] | 42.7 [25.7 to 61.7] | 35.5 [20.4 to 54.0] | 59.8 [40.9 to 76.3] | 52.4 [33.9 to 70.2] | 74.9 [58.0 to 86.6] | 68.7 [50.7 to 82.5]

6. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Peak Forced Expiratory Volume in One Second at Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Peak FEV1 is the maximum FEV1 recorded in a pre-determined period of time.
  Percentage of the maximal response of NVA237 within different doses/regimens of NVA237 on Peak FEV1 was measured at day 28 of treatment.
  Peak FEV1 was measured in response to all doses administered (see Outcome Measure #23). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 82 | 90 | 91 | 89 | 92 | 91 | 82
Percentage of maximal response | 53.3 [41.2 to 65.5] | 69.2 [56.7 to 79.2] | 61.1 [48.2 to 73.4] | 81.5 [71.1 to 88.4] | 75.6 [63.4 to 84.7] | 89.6 [82.4 to 93.9] | 85.8 [76.5 to 91.7]

7. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Vital Capacity at Day 28 of Treatment
Description: Percentage of the maximal response of NVA237 within different doses/regimens of NVA237 on Forced Vital Capacity (FVC) was measured at day 28 of treatment. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
  FVC at day 28 of treatment was measured via spirometry (see Outcome Measure #24). All FVC responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FVC data are reported as a percentage of the theoretical maximal response.
Time Frame: day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 81 | 88 | 90 | 88 | 87 | 90 | 81
Percentage of maximal response | 23.3 [11.3 to 45.3] | 37.4 [19.8 to 62.7] | 53.6 [26.5 to 81.2] | 54.0 [30.9 to 77.2] | 69.3 [38.6 to 89.7] | 69.7 [43.6 to 87.2] | 81.4 [52.5 to 94.6]

8. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Trough Forced Expiratory Volume in One Second at Days 1, 7 and 14
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses on Trough FEV1 was measured on Days 1, 7 and 14.
  Through FEV1 was measured in response to all doses administered (see Outcome Measure #25). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
  Trough FEV1 was defined as the mean of the 23 hour 15 minute and 23 hour 45 minute post-dose values.
Time Frame: Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 88 | 92 | 91 | 91 | 95 | 94 | 87
Percentage of maximal response
  Day 1 (n= 88,92,91, 90, 94, 94, 87) | 28.5 [17.5 to 45.3] | 43.8 [27.8 to 62.3] | 63.3 [37.9 to 82.5] | 60.1 [38.2 to 76.8] | 76.7 [49.3 to 90.5] | 74.3 [48.6 to 86.9] | 86.2 [59.8 to 95.0]
  Day 7 (n= 87,92,90, 91, 95, 93, 85) | 27.1 [16.3 to 44.3] | 42.0 [26.3 to 61.4] | 61.6 [36.4 to 82.1] | 58.5 [37.3 to 76.1] | 75.5 [48.3 to 90.1] | 73.0 [48.7 to 86.4] | 85.4 [59.8 to 94.8]
  Day 14 (n= 85,90,91, 88, 94, 93, 81) | 27.1 [16.4 to 44.3] | 42.0 [26.4 to 61.4] | 61.6 [36.6 to 82.1] | 58.5 [37.4 to 76.1] | 75.5 [48.5 to 90.2] | 73.0 [48.8 to 86.5] | 85.4 [60.1 to 94.8]

9. Secondary Outcome: Percentage of the Maximal Effect of NVA237 Doses on Forced Expiratory Volume in One Second Area Under the Curve 0-24 Hours on Days 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-24 hours, was calculated from measurements taken at 5 min,15 min, 1,2,3,4,6,8,10 hours, 11 hours 55min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on days 1 and 14.
  FEV1 AUC 0-24 hours was measured on days 1 and 14 of treatment in response to all doses administered (see Outcome Measure #26). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 5 min,15 min, 1,2,3,4,6,8,10 hours, 11 hours 55min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on days 1 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87
Percentage of maximal response* hours
  Day 1 (n= 89,94,93,92,96,96,87) | 38.3 [25.3 to 53.4] | 55.4 [40.4 to 69.6] | 59.5 [42.8 to 74.2] | 71.3 [57.5 to 82.1] | 74.6 [60.0 to 85.2] | 83.2 [73.0 to 90.2] | 85.4 [75.0 to 92.0]
  Day 14 (n= 86,92,91,91,95,93,84) | 28.9 [18.7 to 41.6] | 44.8 [31.6 to 58.8] | 49.0 [34.1 to 64.1] | 61.9 [48.0 to 74.0] | 65.7 [50.9 to 78.1] | 76.4 [64.8 to 85.1] | 79.3 [67.5 to 87.7]

10. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second Area Under the Curve 0-4 Hours on Days 1, 7 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer.
  Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-4 hours was calculated from measurements taken at 5 min,15 min, 1,2,3,4 hours (postdose) on Days 1, 7 and 14, in response to all doses administered (see Outcome Measure #27).
  All AUC FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 5 min,15 min, 1,2,3,4 hours (postdose) on Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 86
Percentage of maximal response* hours
  Day 1 (n=89,94,93,91,96,96,86) | 58.4 [44.4 to 71.8] | 73.2 [59.1 to 83.6] | 66.1 [51.6 to 78.6] | 84.1 [72.0 to 91.1] | 79.1 [65.6 to 88.0] | 91.1 [81.5 to 95.3] | 88.0 [77.1 to 93.6]
  Day 7 (n=87,93,90,92,95,94,85) | 50.8 [38.7 to 63.6] | 66.9 [53.7 to 77.7] | 58.9 [45.9 to 71.5] | 79.7 [67.4 to 87.4] | 73.7 [60.6 to 83.4] | 88.3 [77.8 to 93.3] | 84.4 [73.0 to 91.0]
  Day 14 (n=86,92,91,91,95,93,84) | 50.8 [38.7 to 63.6] | 66.9 [53.7 to 77.7] | 58.9 [45.9 to 71.5] | 79.7 [67.4 to 87.4] | 73.7 [60.6 to 83.4] | 88.3 [77.8 to 93.3] | 84.4 [73.0 to 91.0]

11. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second of Area Under the Curve 0-8 Hours Days 1, 7, and 14
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-8 was calculated from measurements taken at 5 min,15 min, 1,2,3,4,6,8 hours (postdose) on days 1, 7, and 14.
  AUC FEV1 was measured in response to all doses administered (see Outcome Measure #28). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: at 5 min,15 min, 1,2,3,4,6,8 hours (postdose) on days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87
Percentage of maximal response* hours
  Day 1 (n=89, 94, 93, 91, 96, 96, 87) | 54.2 [40.1 to 67.8] | 70.3 [57.2 to 80.8] | 63.6 [49.0 to 76.3] | 82.6 [72.8 to 89.4] | 77.8 [65.8 to 86.5] | 90.5 [84.3 to 94.4] | 87.5 [79.4 to 92.8]
  Day 7 (n= 87, 93, 91, 92, 95, 94, 85) | 45.8 [33.2 to 58.8] | 62.8 [49.9 to 74.1] | 55.5 [42.0 to 68.4] | 77.1 [66.6 to 85.1] | 71.4 [59.1 to 81.2] | 87.1 [79.9 to 91.9] | 83.3 [74.3 to 89.7]
  Day 14 (n=86, 92, 91, 91, 95, 93, 84) | 45.8 [33.2 to 58.8] | 62.8 [49.9 to 74.1] | 55.5 [42.0 to 68.4] | 77.1 [66.6 to 85.1] | 71.4 [59.1 to 81.2] | 87.1 [79.9 to 91.9] | 83.3 [74.3 to 89.7]

12. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second Area Under the Curve 0-12 Hours at Day 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses was calculated on FEV1 Area Under the Curve (AUC) 0-12 hours from measurements taken at at 5 min,15 min, 1,2,3,4,6,8,10 hours, 11h 55 min (postdose) on days 1 and 14 in response to all doses administered (see Outcome Measure #29).
  All AUC FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 5 min,15 min, 1,2,3,4,6,8,10 hours, 11h 55 min (postdose) on days 1 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 91 | 96 | 96 | 87
Percentage of maximal response* hours
  Day 1 (n=89, 94, 93, 91, 96, 96, 87) | 49.5 [35.5 to 63.6] | 66.2 [52.4 to 77.8] | 58.8 [44.0 to 72.3] | 79.6 [68.7 to 87.5] | 74.1 [61.1 to 83.9] | 88.7 [81.5 to 93.3] | 85.1 [75.9 to 91.3]
  Day 14 (n=86, 92, 91, 91, 95, 93, 84) | 41.1 [28.8 to 54.5] | 58.3 [44.7 to 70.6] | 50.5 [37.0 to 64.1] | 73.6 [61.8 to 82.8] | 67.1 [54.0 to 78.1] | 84.8 [76.4 to 90.6] | 80.3 [70.1 to 87.7]

13. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second of Area Under the Curve 12-24 Hours Over Days 1, and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 on FEV1 Area under the curve (AUC) 12-24 hours was calculated from measurements taken at 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on Days 1 and 14.
  AUC FEV1 was measured in response to all doses administered (see Outcome Measure #30). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on Days 1 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response* hours
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87
Percentage of maximal response* hours
  Day 1 (n=89, 94, 93, 92, 96, 96, 87) | 23.9 [1.2 to 90.7] | 37.9 [2.4 to 95.2] | 54.4 [4.5 to 97.8] | 54.1 [4.7 to 97.6] | 69.5 [8.6 to 98.9] | 69.3 [9.0 to 98.8] | 81.1 [15.5 to 99.5]
  Day 14 (n= 86, 92, 91, 91, 95, 93, 84) | 25.6 [15.5 to 42.5] | 40.1 [24.2 to 59.6] | 56.6 [31.3 to 78.2] | 56.4 [32.9 to 74.7] | 71.4 [41.4 to 87.8] | 71.2 [42.5 to 85.5] | 82.4 [51.2 to 93.5]

14. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Forced Expiratory Volume in One Second at 12 Hours on Days 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses on FEV1 at 12 hours was measured on days 1 and 14.
  FEV1 was measured in response to all doses administered (see Outcome Measure #31). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: Days 1 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 84 | 91 | 91 | 90 | 90 | 92 | 83
Percentage of maximal response
  Day 1 (n=83, 90, 91, 85, 89, 90, 83) | 35.1 [19.1 to 55.7] | 52.0 [32.0 to 71.6] | 44.4 [25.7 to 64.7] | 68.4 [48.5 to 83.4] | 61.5 [41.0 to 78.5] | 81.2 [65.3 to 91.0] | 76.1 [58.1 to 88.0]
  Day 14 (n=84, 91, 88, 90, 90, 92, 78) | 27.1 [14.7 to 44.6] | 42.7 [25.7 to 61.7] | 35.5 [20.4 to 54.0] | 59.8 [40.9 to 76.3] | 52.4 [33.9 to 70.2] | 74.9 [58.0 to 86.6] | 66.7 [50.7 to 82.5]

15. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Peak Forced Expiratory Volume in One Second on Days 1, 7 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Peak FEV1 is the maximum FEV1 recorded in a pre-determined period of time.
  Percentage of the maximal response of NVA237 doses on Peak FEV1 was measured on days 1, 7 and 14 of treatment.
  Peak FEV1 was measured in response to all doses administered (see Outcome Measure #32). All FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All FEV1 data are reported as a percentage of the theoretical maximal response.
Time Frame: Days 1, 7, and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 86
Percentage of maximal response
  Day 1 (n=89, 94, 93, 91, 96, 96, 86) | 61.7 [47.4 to 74.7] | 76.0 [62.5 to 85.5] | 68.9 [54.1 to 81.1] | 86.1 [75.8 to 92.2] | 81.3 [68.7 to 89.6] | 92.3 [85.6 to 96.0] | 89.5 [80.6 to 94.5]
  Day 7 (n=87, 93, 90, 92, 95, 94, 85) | 53.3 [41.2 to 65.5] | 69.2 [56.7 to 79.2] | 61.1 [48.2 to 73.4] | 81.5 [71.1 to 88.4] | 75.6 [63.4 to 84.7] | 89.6 [82.4 to 93.9] | 85.8 [76.5 to 91.7]
  Day 14 (n=86, 92, 91, 91, 95, 93, 84) | 53.3 [41.2 to 65.5] | 69.2 [56.7 to 79.2] | 61.1 [48.2 to 73.4] | 81.5 [71.1 to 88.4] | 75.6 [63.4 to 84.7] | 89.6 [82.4 to 93.9] | 85.8 [76.5 to 91.7]

16. Secondary Outcome: Percentage of the Maximal Response of NVA237 Doses on Trough Forced Vital Capacity on Days 1, 7 and 14
Description: Percentage of the maximal response of NVA237 Doses on Trough Forced Vital Capacity (FVC) on Days 1, 7 and 14. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FVC was assessed via spirometry. (see Outcome Measure #33).
  Trough FVC is defined as the mean of the FVC values measured at 23 hours 15 mins and 23 hours 45 mins post-dose.
Time Frame: Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 88 | 92 | 91 | 91 | 95 | 94 | 87
Percentage of maximal response
  Day 1 (n=88, 92, 91, 90, 94, 94, 87) | 22.8 [11.3 to 43.5] | 36.8 [19.6 to 60.9] | 52.9 [26.2 to 79.9] | 53.4 [30.7 to 75.8] | 68.7 [38.3 to 88.9] | 69.1 [43.4 to 86.3] | 81.0 [52.3 to 94.1]
  Day 7 (n=87, 92, 90, 91, 95, 93, 85, 87) | 23.3 [11.2 to 45.2] | 37.4 [19.6 to 62.5] | 53.6 [26.3 to 81.2] | 54.0 [30.7 to 77.1] | 69.3 [38.3 to 89.7] | 69.7 [43.3 to 87.1] | 81.4 [52.0 to 94.6]
  Day 14 (n= 85, 90, 91, 88, 94, 93, 81, 84) | 23.3 [11.3 to 45.3] | 37.4 [19.7 to 65.5] | 53.6 [26.4 to 81.2] | 54.0 [30.8 to 77.1] | 69.3 [38.5 to 89.7] | 69.7 [43.5 to 87.2] | 81.4 [52.2 to 94.6]

17. Secondary Outcome: Mean Daily Use of Rescue Medication by Treatment at Different Time Points
Description: Mean daily use of rescue medication by treatment and time points. Baseline was defined as the average of the total number of puffs of rescue medication during the week prior to treatment start, divided by the total number of days with non-missing rescue data during that week, then puffs were counted during weeks 1, 2, 3 and 4 postdose.
Time Frame: Baseline, Weeks 1, 2, 3 and 4
Population: Only patients with a non-missing value at both period baseline and the respective post-baseline visit were included. The modeling approach is not suitable for these data as the modeling assumptions do not hold.
Measure: Mean (Standard Deviation); unit: Number of Puffs
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 95 | 95 | 92 | 96 | 96 | 86 | 91
Number of Puffs
  Baseline (n=89, 95, 95, 92, 96, 96, 86, 91) | 4.16 (3.131) | 4.16 (2.925) | 3.83 (3.218) | 4.45 (3.068) | 3.47 (2.996) | 4.81 (3.276) | 4.25 (3.613) | 4.62 (3.710)
  Week 1 (n=89, 95, 95, 91, 96, 96, 86, 90) | 2.41 (2.338) | 2.23 (2.158) | 2.10 (2.337) | 2.36 (2.291) | 2.13 (2.349) | 2.53 (2.609) | 2.54 (2.678) | 2.94 (3.075)
  Week 2 (n=86, 94, 94, 91, 95, 93, 84, 89) | 2.74 (2.784) | 2.20 (2.054) | 2.22 (2.541) | 2.38 (2.541) | 2.08 (2.568) | 2.59 (2.658) | 2.82 (3.003) | 3.32 (3.455)
  Week 3 (n= 86, 93, 94, 89, 93, 93, 83, 87) | 2.75 (2.736) | 2.40 (2.316) | 2.29 (2.354) | 2.37 (2.580) | 2.23 (2.743) | 2.75 (2.868) | 2.69 (2.977) | 3.34 (3.660)
  Week 4 (n=86, 92, 94, 88, 93, 93, 82, 85) | 2.91 (2.968) | 2.52 (2.476) | 2.42 (2.773) | 2.46 (2.504) | 2.32 (2.990) | 2.65 (2.828) | 2.78 (2.899) | 3.41 (3.761)

18. Primary Outcome: Maximal Response of Incremental Once Daily and Twice Daily Doses of NVA237 That Each Dose Achieves in Relation to the Maximal Effect of NVA237 on Trough Forced Expiratory Volume in One Second at Day 28
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. The maximal response of incremental once daily and twice daily doses of NVA237 that each dose achieves in relation to the maximal effect of NVA237 on Trough FEV1 was measured at Day 28. FEV1 was measured in response to all doses administered (see Outcome Measure #19).
  All trough FEV1 responses to active doses were corrected using the placebo response. A modeled dose response curve was fit to the placebo-corrected data, and extrapolated to estimate the maximal response. All trough FEV1 data are reported as a percentage of the theoretical maximal response.
  Trough FEV1 was defined as the mean of the 23 hour 15 minute and 23 hour 45 minute post-dose values.
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Percentage of maximal response
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d.
Number analyzed (Participants) | 81 | 88 | 90 | 88 | 87 | 90 | 81
Percentage of maximal response | 27.1 (0.454) [16.4 to 44.3] | 42.0 (0.471) [26.5 to 61.4] | 61.6 (0.456) [36.6 to 82.1] | 58.5 (0.389) [37.5 to 76.2] | 75.5 (0.508) [48.7 to 90.2] | 73.0 (0.512) [49.0 to 86.5] | 85.4 (0.463) [60.4 to 94.8]

19. Other Pre Specified Outcome: Trough Forced Expiratory Volume in One Second by Treatment at Day 28
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  Trough FEV1 was defined as the mean of the 23 hour 15 minute and 23 hour 45 minute post-dose values.
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- NVA237 12.5 ug q.d.: NVA237 25 ug once daily
- NVA237 25 ug q.d.: NVA237 12.5 ug once daily
- NVA237 12.5 ug b.i.d.: NVA237 12.5 ug twice daily
- NVA237 50 ug q.d.: NVA237 50 ug once daily
- NVA237 25 ug b.i.d.: NVA237 25 ug twice daily
- NVA237 100 ug q.d.: NVA237 100 ug once daily
- NVA237 50 ug b.i.d.: NVA237 50 ug twice daily
Arm/Group | NVA237 12.5 ug q.d. | NVA237 25 ug q.d. | NVA237 12.5 ug b.i.d. | NVA237 50 ug q.d. | NVA237 25 ug b.i.d. | NVA237 100 ug q.d. | NVA237 50 ug b.i.d. | Placebo
Number analyzed (Participants) | 81 | 88 | 90 | 88 | 87 | 90 | 81 | 82
Liters | 1.319 (0.505) | 1.368 (0.436) | 1.354 (0.484) | 1.340 (0.400) | 1.384 (0.472) | 1.410 (0.522) | 1.493 (0.449) | 1.268 (0.483)

20. Other Pre Specified Outcome: Forced Expiratory Volume in One Second Area Under the Curve 0-24 Hours at Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  FEV1 Area Under the Curve (AUC) measurements were taken at 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on day 28. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 82 | 90 | 91 | 90 | 92 | 91 | 82 | 82
Liters | 1.307 (0.469) | 1.351 (0.392) | 1.321 (0.469) | 1.317 (0.390) | 1.339 (0.462) | 1.395 (0.496) | 1.457 (0.453) | 1.247 (0.467)

21. Other Pre Specified Outcome: Forced Expiratory Volume in One Second Area Under the Curve at Different Time Points (0-4 Hours, 0-8 Hours, 0-12 Hours, 12-24 Hours)
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  FEV1 Area Under the Curve (AUC) measurements were taken at: 5 min,15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose). FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 82 | 90 | 91 | 90 | 92 | 91 | 82 | 82
Liters
  AUC 0-4h (n=82,90,91,89,92,91,82,82) | 1.415 (0.494) | 1.478 (0.439) | 1.414 (0.489) | 1.431 (0.411) | 1.417 (0.487) | 1.490 (0.532) | 1.553 (0.504) | 1.315 (0.490)
  AUC 0-8h (n=82,90,91,90,92,91,82,82) | 1.386 (0.477) | 1.447 (0.423) | 1.392 (0.491) | 1.397 (0.411) | 1.397 (0.476) | 1.461 (0.520) | 1.527 (0.495) | 1.305 (0.485)
  AUC 0-12h (n=82,90,91,90,92,91,82,82) | 1.364 (0.480) | 1.416 (0.416) | 1.362 (0.487) | 1.377 (0.408) | 1.375 (0.469) | 1.442 (0.515) | 1.505 (0.480) | 1.285 (0.476)
  AUC 12-24h (n=82,90,91,89,92,91,81,82) | 1.251 (0.464) | 1.287 (0.382) | 1.280 (0.458) | 1.264 (0.378) | 1.299 (0.459) | 1.350 (0.480) | 1.421 (0.426) | 1.208 (0.461)

22. Other Pre Specified Outcome: Forced Expiratory Volume in One Second at 12 Hours on Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
Time Frame: 12 hours on day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 79 | 88 | 91 | 85 | 87 | 88 | 78 | 80
Liters | 1.272 (0.471) | 1.330 (0.415) | 1.279 (0.476) | 1.330 (0.384) | 1.320 (0.466) | 1.391 (0.498) | 1.429 (0.449) | 1.256 (0.472)

23. Other Pre Specified Outcome: Peak Forced Expiratory Volume in One Second at Day 28 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  Peak FEV1 is the maximum FEV1 recorded in a pre-determined period of time. Measurements were taken at 25 min , 15 min pre-dose, 5 min, 15 min, 1 , 2 ,3 , 4 , 6 , 8 , 10 hours , 11 hour 55 min and 14 hour post-dose on day 28.
Time Frame: 25 min , 15 min pre-dose, 5 min, 15 min, 1 , 2 ,3 , 4 , 6 , 8 , 10 hours , 11 hour 55 min and 14 hour post-dose on day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 82 | 90 | 91 | 89 | 92 | 91 | 82 | 82
Liters | 1.500 (0.516) | 1.563 (0.453) | 1.494 (0.507) | 1.514 (0.432) | 1.504 (0.516) | 1.570 (0.546) | 1.630 (0.513) | 1.397 (0.515)

24. Other Pre Specified Outcome: Trough Forced Vital Capacity After 28 Days of Treatment
Description: Forced Vital Capacity (FVC) after 28 days of treatment. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. Trough FVC was defined as the mean of the FVC values measured at 23 hours 15 mins and 23 hours 45 mins post-dose.
Time Frame: 23 hours 15 mins and 23 hours 45 mins post-dose on Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 81 | 88 | 90 | 88 | 87 | 90 | 81 | 82
Liters | 2.939 (0.878) | 3.007 (0.910) | 2.954 (0.849) | 2.973 (0.825) | 3.041 (0.770) | 2.974 (0.999) | 3.080 (0.913) | 2.703 (0.857)

25. Other Pre Specified Outcome: Trough Forced Expiratory Volume in One Second at Days 1, 7 and 14
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  Trough FEV1 was measured on Days 1, 7 and 14 of treatment. Trough FEV1 was defined as the mean of the FEV1 values measured at 23 hours 15 mins and 23 hours 45 mins post-dose.
Time Frame: 23 hours 15 mins and 23 hours 45 mins post-dose on Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 88 | 92 | 91 | 91 | 95 | 94 | 87 | 87
Liters
  Day 1 (n= 88,92,91, 90, 94, 94, 87, 86) | 1.299 (0.490) | 1.387 (0.477) | 1.375 (0.477) | 1.371 (0.406) | 1.355 (0.503) | 1.367 (0.514) | 1.492 (0.483) | 1.290 (0.471)
  Day 7 (n= 87,92,90, 91, 95, 93, 85, 87) | 1.332 (0.499) | 1.422 (0.432) | 1.349 (0.467) | 1.391 (0.392) | 1.375 (0.486) | 1.372 (0.501) | 1.480 (0.474) | 1.294 (0.491)
  Day 14 (n= 85,90,91, 88, 94, 93, 81, 84) | 1.336 (0.442) | 1.349 (0.446) | 1.335 (0.444) | 1.356 (0.391) | 1.359 (0.479) | 1.375 (0.519) | 1.500 (0.455) | 1.284 (0.471)

26. Other Pre Specified Outcome: Forced Expiratory Volume in One Second Area Under the Curve 0-24 Hours on Days 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  FEV1 Area Under the Curve (AUC) measurements were taken at 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on days 1 and 14 of treatment. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 5 min, 15 min, 1,2,3,4,6,8,10 hours, 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on days 1 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87 | 90
Liters
  Day 1 (n= 89,94,93,92,96,96,87,90) | 1.318 (0.470) | 1.370 (0.444) | 1.354 (0.462) | 1.361 (0.393) | 1.336 (0.460) | 1.376 (0.526) | 1.466 (0.471) | 1.256 (0.469)
  Day 14 (n= 86,92,91,91,95,93,84,86) | 1.306 (0.427) | 1.353 (0.420) | 1.324 (0.430) | 1.348 (0.372) | 1.335 (0.460) | 1.386 (0.493) | 1.449 (0.453) | 1.253 (0.473)

27. Other Pre Specified Outcome: Forced Expiratory Volume in One Second Area Under the Curve 0-4 Hours on Days 1, 7 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Spirometry was performed according to internationally accepted standards.
  FEV1 Area Under the Curve (AUC) measurements were taken at 5 min, 15 min, 1,2,3,4 hours (postdose) on days 1, 7 and 14 of treatment. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 5 min,15 min, 1,2,3,4 hours (postdose) on Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 86 | 89
Liters
  Day 1 (n=89,94,93,91,96,96,86,89) | 1.428 (0.492) | 1.483 (0.485) | 1.421 (0.489) | 1.469 (0.428) | 1.411 (0.483) | 1.453 (0.551) | 1.533 (0.501) | 1.312 (0.494)
  Day 7 (n=87,93,90,92,95,94,85,89) | 1.403 (0.468) | 1.483 (0.463) | 1.397 (0.478) | 1.432 (0.407) | 1.390 (0.472) | 1.453 (0.505) | 1.537 (0.494) | 1.310 (0.491)
  Day 14 (n=86,92,91,91,95,93,84,86) | 1.451 (0.456) | 1.473 (0.456) | 1.390 (0.471) | 1.468 (0.409) | 1.429 (0.503) | 1.460 (0.514) | 1.545 (0.485) | 1.314 (0.500)

28. Other Pre Specified Outcome: Forced Expiratory Volume in One Second of Area Under the Curve 0-8 Hours Days 1, 7, and 14
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses on FEV1 Area Under the Curve (AUC) 0-8 was calculated from measurements taken at 5 min,15 min, 1,2,3,4,6,8 hours (postdose) on days 1, 7, and 14. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: at 5 min,15 min, 1,2,3,4,6,8 hours (postdose) on days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87 | 90
Liters
  Day 1 (n=89, 94, 93, 91, 96, 96, 87, 90) | 1.400 (0.486) | 1.450 (0.476) | 1.401 (0.483) | 1.451 (0.426) | 1.390 (0.476) | 1.446 (0.548) | 1.519 (0.493) | 1.301 (0.488)
  Day 7 (n= 87, 93, 91, 92, 95, 94, 85, 89) | 1.386 (0.471) | 1.462 (0.455) | 1.375 (0.464) | 1.409 (0.397) | 1.373 (0.470) | 1.433 (0.503) | 1.516 (0.481) | 1.293 (0.489)
  Day 14 (n=86, 92, 91, 91, 95, 93, 84, 86) | 1.381 (0.453) | 1.441 (0.452) | 1.375 (0.463) | 1.435 (0.398) | 1.400 (0.486) | 1.442 (0.508) | 1.514 (0.479) | 1.293 (0.498)

29. Other Pre Specified Outcome: Forced Expiratory Volume in One Second Area Under the Curve 0-12 Hours at Day 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses was calculated on FEV1 Area Under the Curve (AUC) 0-12 hours from measurements taken at at 5 min,15 min, 1,2,3,4,6,8,10 hours, 11h 55 min (postdose) on days 1 and 14. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 5 min,15 min, 1,2,3,4,6,8,10 hours, 11h 55 min (postdose) on days 1 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 91 | 96 | 96 | 87 | 90
Liters
  Day 1 (n=89, 94, 93, 91, 96, 96, 87, 90) | 1.382 (0.488) | 1.425 (0.465) | 1.379 (0.474) | 1.430 (0.421) | 1.364 (0.470) | 1.431 (0.544) | 1.498 (0.484) | 1.289 (0.482)
  Day 14 (n=86, 92, 91, 91, 95, 93, 84, 86) | 1.360 (0.447) | 1.416 (0.445) | 1.357 (0.452) | 1.406 (0.388) | 1.378 (0.480) | 1.427 (0.503) | 1.494 (0.472) | 1.281 (0.493)

30. Other Pre Specified Outcome: Forced Expiratory Volume in One Second of Area Under the Curve 12-24 Hours Over Days 1, and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 on FEV1 Area under the curve (AUC) 12-24 hours was calculated from measurements taken at 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on Days 1 and 14. FEV1 AUC was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 11 hours 55 min, 14,20,22 hours; 23 hours 15 min, 23 hours 45 min (postdose) on Days 1 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 87 | 90
Liters
  Day 1 (n=89, 94, 93, 92, 96, 96, 87, 90) | 1.257 (0.459) | 1.315 (0.432) | 1.329 (0.455) | 1.295 (0.375) | 1.306 (0.454) | 1.322 (0.512) | 1.437 (0.461) | 1.224 (0.459)
  Day 14 (n= 86, 92, 91, 91, 95, 93, 84, 86) | 1.251 (0.417) | 1.289 (0.405) | 1.290 (0.415) | 1.291 (0.366) | 1.291 (0.450) | 1.344 (0.488) | 1.406 (0.437) | 1.225 (0.459)

31. Other Pre Specified Outcome: Forced Expiratory Volume in One Second at 12 Hours on Days 1 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Percentage of the maximal response of NVA237 doses on FEV1 at 12 hours was measured on days 1 and 14.
Time Frame: Days 1 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 84 | 91 | 91 | 90 | 90 | 92 | 83 | 83
Liters
  Day 1 (n=83, 90, 91, 85, 89, 90, 83, 81) | 1.319 (0.502) | 1.364 (0.452) | 1.327 (0.465) | 1.345 (0.405) | 1.299 (0.457) | 1.374 (0.549) | 1.439 (0.459) | 1.244 (0.449)
  Day 14 (n=84, 91, 88, 90, 90, 92, 78, 83) | 1.290 (0.431) | 1.356 (0.431) | 1.303 (0.428) | 1.329 (0.368) | 1.329 (0.455) | 1.389 (0.506) | 1.469 (0.436) | 1.268 (0.477)

32. Other Pre Specified Outcome: Peak Forced Expiratory Volume in One Second on Days 1, 7 and 14 of Treatment
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Peak FEV1 is the maximum FEV1 recorded in a pre-determined period of time.
  Percentage of the maximal response of NVA237 doses on Peak FEV1 was measured on days 1, 7 and 14 of treatment.
Time Frame: Days 1, 7, and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 89 | 94 | 93 | 92 | 96 | 96 | 86 | 89
Liters
  Day 1 (n=89, 94, 93, 91, 96, 96, 86, 89) | 1.503 (0.515) | 1.558 (0.497) | 1.494 (0.507) | 1.541 (0.442) | 1.483 (0.495) | 1.521 (0.567) | 1.597 (0.510) | 1.378 (0.504)
  Day 7 (n=87, 93, 90, 92, 95, 94, 85, 89) | 1.459 (0.477) | 1.540 (0.474) | 1.455 (0.496) | 1.501 (0.426) | 1.448 (0.491) | 1.513 (0.524) | 1.598 (0.510) | 1.364 (0.504)
  Day 14 (n=86, 92, 91, 91, 95, 93, 84, 86) | 1.487 (0.471) | 1.547 (0.465) | 1.465 (0.484) | 1.537 (0.429) | 1.506 (0.513) | 1.528 (0.529) | 1.615 (0.497) | 1.380 (0.509)

33. Other Pre Specified Outcome: Trough Forced Vital Capacity on Days 1, 7 and 14
Description: Trough Forced Vital Capacity (FVC) on Days 1, 7 and 14. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. (see Outcome Measure #23).
  Trough FVC was defined as the mean of the 23 hour 15 minute and 23 hour 45 minute post-dose values.
Time Frame: Days 1, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 12.5 µg q.d. | NVA237 25.0 µg q.d. | NVA237 12.5 µg b.i.d. | NVA237 50.0 µg q.d. | NVA237 25.0 µg b.i.d. | NVA237 100.0 µg q.d. | NVA237 50.0 µg b.i.d. | Placebo
Number analyzed (Participants) | 88 | 92 | 91 | 91 | 95 | 94 | 87 | 87
Liters
  Day 1 (n=88, 92, 91, 90, 94, 94, 87, 86) | 2.895 (0.830) | 3.063 (0.967) | 2.997 (0.835) | 3.017 (0.820) | 2.956 (0.810) | 2.944 (1.001) | 3.088 (0.961) | 2.779 (0.838)
  Day 7 (n=87, 92, 90, 91, 95, 93, 85, 87) | 2.982 (0.833) | 3.135 (0.928) | 2.991 (0.873) | 3.072 (0.833) | 2.993 (0.798) | 2.977 (0.987) | 3.114 (0.975) | 2.759 (0.875)
  Day 14 (n= 85, 90, 91, 88, 94, 93, 81, 84) | 2.958 (0.772) | 3.000 (0.934) | 2.965 (0.862) | 3.003 (0.812) | 2.960 (0.763) | 2.941 (0.987) | 3.113 (0.941) | 2.744 (0.841)

ADVERSE EVENTS:
Groups:
- NVA237 12.5 ug q.d.: NVA237 12.5 ug q.d.
- NVA237 25 ug q.d.: NVA237 25 ug q.d.
- NVA237 12.5 ug b.i.d.: NVA237 12.5 ug b.i.d.
- NVA237 50 ug q.d.: NVA237 50 ug q.d.
- NVA237 25 ug b.i.d.: NVA237 25 ug b.i.d.
- NVA237 100 ug q.d.: NVA237 100 ug q.d.
- NVA237 50 ug b.i.d.: NVA237 50 ug b.i.d.
- Placebo: Placebo
Arm/Group | NVA237 12.5 ug q.d. | NVA237 25 ug q.d. | NVA237 12.5 ug b.i.d. | NVA237 50 ug q.d. | NVA237 25 ug b.i.d. | NVA237 100 ug q.d. | NVA237 50 ug b.i.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 2/89 | 2/96 | 1/96 | 3/92 | 4/96 | 3/96 | 1/87 | 3/91
Other Adverse Events (participants affected / at risk) | 9/89 | 11/96 | 5/96 | 7/92 | 8/96 | 9/96 | 9/87 | 14/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 12.5 ug q.d. (N=89) | NVA237 25 ug q.d. (N=96) | NVA237 12.5 ug b.i.d. (N=96) | NVA237 50 ug q.d. (N=92) | NVA237 25 ug b.i.d. (N=96) | NVA237 100 ug q.d. (N=96) | NVA237 50 ug b.i.d. (N=87) | Placebo (N=91)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 12.5 ug q.d. (N=89) | NVA237 25 ug q.d. (N=96) | NVA237 12.5 ug b.i.d. (N=96) | NVA237 50 ug q.d. (N=92) | NVA237 25 ug b.i.d. (N=96) | NVA237 100 ug q.d. (N=96) | NVA237 50 ug b.i.d. (N=87) | Placebo (N=91)
Nasopharyngitis (Infections and infestations) | 4 | 8 | 2 | 4 | 3 | 4 | 5 | 6
Headache (Nervous system disorders) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1 | 0 | 3 | 2 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.